CLINICAL TRIAL: NCT00221143
Title: Phase I / II Clinical Trial Regarding Vascular Regeneration Therapy by Transplantation of Autologous Peripheral Blood Endothelial Progenitor Cells (CD34+ Cells) in No-Option Patients With Chronic Critical Limb Ischemia
Brief Title: Stem Cell Study for Patients With Leg Ulcer/Gangrene
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Institute of Biomedical Research and Innovation, Kobe, Hyogo, Japan (Other); Kobe City General Hospital (Other)
Responsible Party: Atsuhiko Kawamoto, MD, PhD Senior Research Scientist, Stem Cell Translational research Team, Institute of Biomedical Research and Innovation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRI ASO 03-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-02

CONDITIONS: Leg Pain; Ulcer; Gangrene; Ischemia; Peripheral Vascular Diseases
Keywords: Ulcer/ gangrene; Leg diseases; Pain; Vascular diseases; Chronic limb ischemia; Peripheral artery disease
MeSH Terms: conditions — Ulcer; Gangrene; Ischemia; Peripheral Vascular Diseases; Pain; Vascular Diseases; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: Autologous peripheral blood CD34 positive cell therapy

SUMMARY:
The purpose of this study is to determine if stem cell therapy with one's own cells (autologous cells) delivered intramuscularly to one's leg with ulcer and/or gangrene due to poor blood flow will be safe and if it will relieve leg pain, increase blood flow, and/or cure the leg wound.

DETAILED DESCRIPTION:
Chronic critical limb ischemia (CLI) is a progressive disease, which arises as a result of atherosclerosis or vasculitis in leg arteries. Prognosis of chronic CLI is poor, and no effective treatments have been established in patients who are not eligible for the traditional revascularization therapies such as angioplasty and bypass procedures due to the inappropriate anatomy of the leg arteries or frequent reocclusion following revascularization. Therefore, it is necessary to establish novel revascularization treatment to improve prognosis of the no-option patients. We will study the safety and clinical efficiency of vascular regeneration by means of transplantation of autologous peripheral blood endothelial progenitor cells (CD34 positive cells) in patients with chronic CLI who are not eligible for traditional revascularization treatments. The primary endpoint is the primary efficacy score identified by toe brachial blood pressure index (TBPI), absolute claudication distance (ACD) and Wong Baker's pain rating scale, while the secondary endpoints are evaluation of safety, ankle brachial blood pressure index (ABPI), percutaneous tissue oxygen pressure (TcPO2), etc.

ELIGIBILITY:
Inclusion Criteria:

* Chronic severe CLI patients fulfilling all the following criteria are considered suitable for inclusion in the study.

  1. At least 6 months since the onset of CLI (Chronic peripheral artery disease or Buerger disease)
  2. Patients with luminal stenosis > 50% by leg angiography
  3. Age is between 20 and 80.
  4. Patients whose Rutherford's class is II-4, III-5, or III-6（Patients with rest pain or ischemic ulcer/necrosis)
  5. Patients for whom angioplasty and bypass surgery are not indicated because of anatomical or procedural reasons or frequent reocclusion/ restenosis following the traditional revascularization (No option patients)
  6. Patients who can give informed consent themselves in writing.

Exclusion Criteria:

* Any one of the following exclusion criteria is sufficient to disqualify a patient from the study.

  1. Left ventricular ejection fraction < 25%
  2. Patients with a history of severe allergic reactions or side effects to G-CSF preparations or apheresis.
  3. Less than 6 months since last episode of myocardial/cerebral infarction.
  4. Patients with unstable angina, with a treatment rating of 3 in the Braunwald system, but a severity of III and a clinical rating of B or C.
  5. Patients with diabetic proliferating retinopathy (new Fukuda classification BI to BV).
  6. Patients with malignant tumor
  7. Patients with chronic rheumatoid arthritis.
  8. Patients with hematological disease (leukemia, myeloproliferative disease, or myelodysplastic syndromes).
  9. Patients currently suffering from or having a history of interstitial pneumonitis.
  10. Patients for whom cranial MRA reveals cerebral aneurysm.
  11. Patients for whom abdominal CT or ultrasonography reveals splenomegaly.
  12. Patients with cirrhosis of the liver.
  13. Patients who cannot discontinue Warfarin.
  14. Leukocytes less than 4,000/µL or exceeding 10,000/µL.
  15. Platelets less than 100,000/µL.
  16. Hemoglobin less than 10 g/dL.
  17. AST (GOT) exceeding 100 IU/L or ALT (GPT) exceeding 100 IU/L.
  18. Patients with severe neural disorder in their legs.
  19. Patients with gait disturbance for reasons other than CLI (such as sciatic neuralgia, or vasculitis), making exercise tolerance evaluation on a treadmill with stress ECG difficult.
  20. Pregnant or nursing patients, those who may be pregnant, or those who plan on becoming pregnant before the end of the study period.
  21. Any other reason that the Clinical Supervisors or Clinical Researchers may have for considering a case unsuitable for the study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-11; Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Major amputation

SECONDARY OUTCOMES:
Limb ischemia

CONTACTS AND LOCATIONS:
Overall Officials: Takayuki Asahara, M.D., Principal Investigator — Institute of Biomedical Research and Innovation, Kobe, Hyogo, Japan
Locations (2):
- Japan (2):
  - Kobe City General Hospital, Kobe, Hyōgo
  - Institute of Biomedical Research and Innovation, Kobe, Hyōgo

REFERENCES:
- [Background] Asahara T, Kawamoto A. Endothelial progenitor cells for postnatal vasculogenesis. Am J Physiol Cell Physiol. 2004 Sep;287(3):C572-9. doi: 10.1152/ajpcell.00330.2003. PMID 15308462
- [Background] Kawamoto A, Tkebuchava T, Yamaguchi J, Nishimura H, Yoon YS, Milliken C, Uchida S, Masuo O, Iwaguro H, Ma H, Hanley A, Silver M, Kearney M, Losordo DW, Isner JM, Asahara T. Intramyocardial transplantation of autologous endothelial progenitor cells for therapeutic neovascularization of myocardial ischemia. Circulation. 2003 Jan 28;107(3):461-8. doi: 10.1161/01.cir.0000046450.89986.50. PMID 12551872
- [Background] Kawamoto A, Gwon HC, Iwaguro H, Yamaguchi JI, Uchida S, Masuda H, Silver M, Ma H, Kearney M, Isner JM, Asahara T. Therapeutic potential of ex vivo expanded endothelial progenitor cells for myocardial ischemia. Circulation. 2001 Feb 6;103(5):634-7. doi: 10.1161/01.cir.103.5.634. PMID 11156872
- [Background] Asahara T, Murohara T, Sullivan A, Silver M, van der Zee R, Li T, Witzenbichler B, Schatteman G, Isner JM. Isolation of putative progenitor endothelial cells for angiogenesis. Science. 1997 Feb 14;275(5302):964-7. doi: 10.1126/science.275.5302.964. PMID 9020076
- [Background] Takahashi T, Kalka C, Masuda H, Chen D, Silver M, Kearney M, Magner M, Isner JM, Asahara T. Ischemia- and cytokine-induced mobilization of bone marrow-derived endothelial progenitor cells for neovascularization. Nat Med. 1999 Apr;5(4):434-8. doi: 10.1038/7434. PMID 10202935
- [Background] Kalka C, Masuda H, Takahashi T, Kalka-Moll WM, Silver M, Kearney M, Li T, Isner JM, Asahara T. Transplantation of ex vivo expanded endothelial progenitor cells for therapeutic neovascularization. Proc Natl Acad Sci U S A. 2000 Mar 28;97(7):3422-7. doi: 10.1073/pnas.97.7.3422. PMID 10725398
- [Derived] Kinoshita M, Fujita Y, Katayama M, Baba R, Shibakawa M, Yoshikawa K, Katakami N, Furukawa Y, Tsukie T, Nagano T, Kurimoto Y, Yamasaki K, Handa N, Okada Y, Kuronaka K, Nagata Y, Matsubara Y, Fukushima M, Asahara T, Kawamoto A. Long-term clinical outcome after intramuscular transplantation of granulocyte colony stimulating factor-mobilized CD34 positive cells in patients with critical limb ischemia. Atherosclerosis. 2012 Oct;224(2):440-5. doi: 10.1016/j.atherosclerosis.2012.07.031. Epub 2012 Jul 27. PMID 22877866
- [Derived] Kawamoto A, Katayama M, Handa N, Kinoshita M, Takano H, Horii M, Sadamoto K, Yokoyama A, Yamanaka T, Onodera R, Kuroda A, Baba R, Kaneko Y, Tsukie T, Kurimoto Y, Okada Y, Kihara Y, Morioka S, Fukushima M, Asahara T. Intramuscular transplantation of G-CSF-mobilized CD34(+) cells in patients with critical limb ischemia: a phase I/IIa, multicenter, single-blinded, dose-escalation clinical trial. Stem Cells. 2009 Nov;27(11):2857-64. doi: 10.1002/stem.207. PMID 19711453